CLINICAL TRIAL: NCT04333810
Title: Remote Physiologic Monitoring to Detect Inflammatory Bowel Disease (IBD) Flares: A Feasibility Study
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Tinsley, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY14888
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Remote monitoring; Heart rate variability; Whoop strap 3.0
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active IBD patients: Patients with active IBD, based on colonoscopic evaluation and biopsy results.
  Interventions: Device: Whoop strap 3.0
- IBD patients in remission: IBD patients in remission, with no recently colonoscopic evidence of disease, and only on maintenance therapy.
  Interventions: Device: Whoop strap 3.0

INTERVENTIONS:
Device: Whoop strap 3.0 — WHOOP strap 3.0, a photodiode-based device that tracks sleep duration, resting heart rate, heart rate variability, activity (calories).

SUMMARY:
Inflammatory bowel disease (IBD) has become a more prominent disease in the US population, with more than 3 million adults in the US affected. To manage this disease effectively, physicians tend to need to have a multidisciplinary approach as there are many psychosocial implications of chronic gastrointestinal illnesses like Crohn's and Ulcerative Colitis. Recent literature has supported the desire for telemedicine and remote physiologic monitoring for such patients to allow the patient to be more active in their treatments and make physicians more aware of what their bodies are doing from a physiologic perspective. Whoop is a new device founded in 2011 that has grown in popularity for its ability to accurately measure sleep patterns, resting heart rate, and heart rate variability (HRV) amongst other various physiologic measurements. Newer literature supports that depressed heart rate variability can correlate to disease flares such as heart failure exacerbations. The study investigators proposed that using remote physiologic monitoring in the IBD population along with their symptoms can help predict disease severity and potentially lead to earlier interventions if correlations are accurate. It can also spark interest in the younger generation for remote physiologic monitoring and telemedicine, which is believed to be beneficial in patients with chronic illnesses.

DETAILED DESCRIPTION:
The prevalence of inflammatory bowel disease continues to rise in the United States, with an estimated 3 million adults carrying this diagnosis in 2015. With inflammatory bowel disease (IBD) comes significant psychosocial implications [Carson, 2013].These patients often feel alone and isolated due to their underlying disease burden. Literature has supported that subjectively; these patients often feel like they are isolated and also have a poor quality of life [Jones, 2019]. One of the biggest factors that has been evaluated in determining quality of life has been sleep. With the aid of the Pittsburgh Quality Sleep Index (PSQI), there has been proof that patients with active disease have poor sleep quality compared to their counterparts with IBD patients in general having worse sleep cycles as compared to healthy individuals [Sobolewska-Wlodarczyk, 2018; Ananthakrishnan, 2013]. It is hypothesized that disruption of the circadian system increases the release of inflammatory cytokines and immune activation, playing a role in chronic inflammatory diseases [Swanson, 2011]. Despite these correlations with sleep via subjective measures, no great objective data has been collected on this patient population.

Another physiologic measurement that has been used for prediction and management of chronic diseases is heart rate variability (HRV). One highly investigated disease was heart failure [Jimenez-Morgan, 2017; Goessl, 2017, Shaffer, 2017; Bullinga; 2005; Tsuji, 1996]. The metric of HRV was used to predict mortality in heart failure with reduced ejection fraction and new cardiac events for which depressed HRV was predictive of more disease burden [Liu, 2014]. Other chronic diseases have yet been explored in regard to quantifiable physiologic measures.

There has been a push amongst all providers to search for a better way to connect with their patients. Multiple mobile applications have been explored, especially in the IBD community [Riaz, 2016]. These individuals are wanting to be more involved in their care and be kept in the loop. The investigators propose utilizing the Whoop Strap 3.0 to evaluate a number of physiologic metrics as well as sleep measures. Telemonitoring is currently being explored in this population, but there is a desire for something more that can quantify data: remote physiologic monitoring. This device can also help with shared decision making and have the patient directly involved in his or her care [Baars, 2010]. A recent study validated the Whoop device for sleep tracking and compared it to polysomnography, nearly identical in their results [Berryhill, 2020]. The device can also promote good healthy lifestyles with exercise, which is known to beneficial in this population [Engels, 2017].

For this project, the investigators propose to investigate disease activity in accordance to physiologic and lifestyle measures utilizing the Whoop strap 3.0. This device and mobile application allow the patient to input everyday symptoms and overall activity which can allow us to correlate some subjective symptoms of potential disease flare with physiologic measurements. There is no published literature looking at the IBD population and has only been investigated in the cardiology realm, which has shown some positive correlation with chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients at Penn State Milton S. Hershey Medical Center
* Age greater than 18

Exclusion Criteria:

* Inability to wear Whoop Strap 3.0 for 24 hours per day for 6 months
* Subjects who are pregnant
* Subjects who are on anti-arrhythmic medications
* Subjects who are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inflammatory Bowel Disease (IBD) patients at Penn State Milton S. Hershey Medical Center with either active disease or inactive disease (remission) will be enrolled in this study according to the inclusion and exclusion criteria below.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease flares | 6 months
  Inflammatory Bowel Disease flares will be assessed by symptomatology and verified by colonoscopic biopsies to confirm active disease, reemergence of disease, or new disease.
Change in Sleep (hours per night) | 6 months, change measured every 2 weeks
  Sleep will be objectively measured nightly using the wearable Whoop strap 3.0, and averages will be compared every 2 weeks over the duration of the study.
Change in Heart Rate Variability (HRV) | 6 months, change measured every 2 weeks
  Heart Rate Variability will be objectively measured nightly using the wearable Whoop strap 3.0. Average two-week values will be assessed for change every 2 weeks over the duration of the study.
Change in Resting Heart Rate (RHR) | 6 months, change measured every 2 weeks
  Resting Heart Rate will be objectively measured nightly using the wearable Whoop strap 3.0. Average two-week values will be assessed for change every 2 weeks over the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tinsley, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carson HJ, Dudley MH, Knight LD, Lingamfelter D. Psychosocial complications of Crohn's disease and cause of death. J Forensic Sci. 2014 Mar;59(2):568-70. doi: 10.1111/1556-4029.12314. PMID 24749148
- [Background] Jones JL, Nguyen GC, Benchimol EI, Bernstein CN, Bitton A, Kaplan GG, Murthy SK, Lee K, Cooke-Lauder J, Otley AR. The Impact of Inflammatory Bowel Disease in Canada 2018: Quality of Life. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S42-S48. doi: 10.1093/jcag/gwy048. Epub 2018 Nov 2. PMID 31294384
- [Background] Sobolewska-Wlodarczyk A, Wlodarczyk M, Banasik J, Gasiorowska A, Wisniewska-Jarosinska M, Fichna J. Sleep disturbance and disease activity in adult patients with inflammatory bowel diseases. J Physiol Pharmacol. 2018 Jun;69(3). doi: 10.26402/jpp.2018.3.09. Epub 2018 Sep 28. PMID 30279306
- [Background] Ananthakrishnan AN, Long MD, Martin CF, Sandler RS, Kappelman MD. Sleep disturbance and risk of active disease in patients with Crohn's disease and ulcerative colitis. Clin Gastroenterol Hepatol. 2013 Aug;11(8):965-71. doi: 10.1016/j.cgh.2013.01.021. Epub 2013 Feb 1. PMID 23376797
- [Background] Swanson GR, Gorenz A, Shaikh M, Desai V, Forsyth C, Fogg L, Burgess HJ, Keshavarzian A. Decreased melatonin secretion is associated with increased intestinal permeability and marker of endotoxemia in alcoholics. Am J Physiol Gastrointest Liver Physiol. 2015 Jun 15;308(12):G1004-11. doi: 10.1152/ajpgi.00002.2015. Epub 2015 Apr 23. PMID 25907689
- [Background] Jimenez Morgan S, Molina Mora JA. Effect of Heart Rate Variability Biofeedback on Sport Performance, a Systematic Review. Appl Psychophysiol Biofeedback. 2017 Sep;42(3):235-245. doi: 10.1007/s10484-017-9364-2. PMID 28573597
- [Background] Goessl VC, Curtiss JE, Hofmann SG. The effect of heart rate variability biofeedback training on stress and anxiety: a meta-analysis. Psychol Med. 2017 Nov;47(15):2578-2586. doi: 10.1017/S0033291717001003. Epub 2017 May 8. PMID 28478782
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Bullinga JR, Alharethi R, Schram MS, Bristow MR, Gilbert EM. Changes in heart rate variability are correlated to hemodynamic improvement with chronic CARVEDILOL therapy in heart failure. J Card Fail. 2005 Dec;11(9):693-9. doi: 10.1016/j.cardfail.2005.06.435. PMID 16360965
- [Background] Tsuji H, Larson MG, Venditti FJ Jr, Manders ES, Evans JC, Feldman CL, Levy D. Impact of reduced heart rate variability on risk for cardiac events. The Framingham Heart Study. Circulation. 1996 Dec 1;94(11):2850-5. doi: 10.1161/01.cir.94.11.2850. PMID 8941112
- [Background] Liu G, Wang L, Wang Q, Zhou G, Wang Y, Jiang Q. A new approach to detect congestive heart failure using short-term heart rate variability measures. PLoS One. 2014 Apr 18;9(4):e93399. doi: 10.1371/journal.pone.0093399. eCollection 2014. PMID 24747432
- [Background] Riaz MS, Atreja A. Personalized Technologies in Chronic Gastrointestinal Disorders: Self-monitoring and Remote Sensor Technologies. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1697-1705. doi: 10.1016/j.cgh.2016.05.009. Epub 2016 May 14. PMID 27189911
- [Background] Baars JE, Markus T, Kuipers EJ, van der Woude CJ. Patients' preferences regarding shared decision-making in the treatment of inflammatory bowel disease: results from a patient-empowerment study. Digestion. 2010;81(2):113-9. doi: 10.1159/000253862. Epub 2010 Jan 9. PMID 20093836
- [Background] Berryhill S, Morton CJ, Dean A, Berryhill A, Provencio-Dean N, Patel SI, Estep L, Combs D, Mashaqi S, Gerald LB, Krishnan JA, Parthasarathy S. Effect of wearables on sleep in healthy individuals: a randomized crossover trial and validation study. J Clin Sleep Med. 2020 May 15;16(5):775-783. doi: 10.5664/jcsm.8356. Epub 2020 Feb 11. PMID 32043961
- [Background] Engels M, Cross RK, Long MD. Exercise in patients with inflammatory bowel diseases: current perspectives. Clin Exp Gastroenterol. 2017 Dec 22;11:1-11. doi: 10.2147/CEG.S120816. eCollection 2018. PMID 29317842